CLINICAL TRIAL: NCT06995716
Title: Assessment Of Spinal Posture, Balance And Ankle Muscle Shortness İn Children With Autism
Status: Enrolling by invitation | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Seda AYAZ TAŞ, Assistant Professor Dr., Abant Izzet Baysal University
Other Study IDs: BAIBU-FTR-SAT-9
Record Dates: First submitted 2025-05-21; First posted 2025-05-29 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Typically Developing Children: This group consists of typically developing children.
- Children With Autism: This group consists of children who have been diagnosed with autism based on "Special Needs Report for Children" (ÇÖZGER) report.

SUMMARY:
The aim of this study is to evaluate spinal posture, mobility, balance and ankle muscle shortness in children with autism.

The study will feature two groups,

* First group will consist of children with autism
* Second group will consist of typically developing children

Childhood autism assessment scale will be completed with the families of the children included in the study. The tiptoe walking status of the children participating in the study will be observed and classified according to the tiptoe walking classification. Children's balance skills will be evaluated with pediatric berg balance test and timed get up and walk test, ankle muscle shortness will be evaluated with Gastro-Soleus shortness measurements, spinal posture and mobility will be evaluated with spinal mouse.

The evaluation results of both groups will be compared.

The main questions this study aims to answer are:

* Is spinal mobility decreased in children with autism compared to typically developing children?
* Is Thoracic kyphosis greater in children with autism compared to typically developing children?
* Are Balance skills poorer in children with autism compared to typically developing children?
* Does the severity of tiptoe walking increase as gastro-soleus muscle shortness increases?

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with autism spectrum disorder in the Special Needs Report for Children (ÇÖZGER)
* GMFCS level I or II
* Between the ages of 6-18
* IQ score of 50 or more as determined in the Special Needs Report for Children (ÇÖZGER)
* Volunteering to participate in the study

Exclusion Criteria:

* Having a rigid contracture of the columna vertebralis
* Having undergone scoliosis surgery
* Having a rigid contracture in passive knee extension and ankle range of motion
* History of surgery or botox affecting ankle joint range of motion in the last 6 months

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: This study includes children with autism and typically developing children between the ages of 6-18
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
Spinal posture and mobility | 6 Months
  Spinal Mouse :
  Spinal Mouse is a tool used for noninvasive external evaluation that measures spinal angles and shape in frontal and sagittal planes. It is used to measure spinal intersegmental angles and spinal range of motion. The device is moved over the columna vertebralis on the skin surface following the spinous processes from C7 to S3. It provides information about inclination, thorax, lumbar and sacrum/hip angles. Stores data and provides result output via computer program
  Both frontal and sagittal assesment were made while standing upright
  For the sagittal assesment there were 3 different evaluation positions
  * Standing still
  * Body flexion
  * Body extension
  For the frontal assesment there were 3 different evaluation positions
  * Standing still
  * Body left lateral flexion
  * Body right lateral flexion

SECONDARY OUTCOMES:
Childhood Autism Rating Scale | 6 Months
  It is a scale consisting of 15 items used to assess the severity of autism, with each item scored between 1 and 4. A score of 1 represents that the child's behavior for that item is normal for his/her age, while a score of 4 represents that it is extremely abnormal. The minimum score is 15 and the maximum score is 60. The results are evaluated as "no autism" between 15-29 points, "mild-moderate autism" between 30-36 points, and extreme autism between 37-60 points.
  Families of the children were asked to fill out the forms.
Pediatric Berg Balance Scale | 6 Months
  It is a scale used to assess the balance of 14 functional tasks. Each item is scored between 0 and 4. A higher score represents better balance. The maximum possible score is 56.
  Children were asked to complete the functional tasks and were scored accordingly to their performance.
Timed Up and Go Test | 6 Months
  Children were asked to sit upright on a chair with a straight back. At the start command, the child stood up, walked 3 meters, turned around and sat back on the chair. The time taken to perform the movement was recorded in seconds and performance was interpreted accordingly
M.Gastrocnemius - M.Gastrosoleus Shortness Measurement | 6 Months
  Passive foot dorsiflexion measurement with a manual goniometer was performed at 0 degrees knee flexion for Gastrocnemius muscle and 90 degrees knee flexion for Soleus muscle. Muscle shortness was expressed in degrees. Ankle neutral position was recorded as 0 degrees, dorsiflexion angles as positive and plantar flexion angles as negative.
Classification of Tiptoe Walking | 6 Months
  Tiptoe walking was assessed and classified by observation during 10-meter walk-run. Level 1 indicates that there is tiptoe behavior during running, walking and standing; Level 2 indicates that there is tiptoe behavior during running and walking; Level 3 indicates that there is tiptoe behavior only during running; if no tiptoe walking is observed, it was indicated as "no tiptoe walking".

CONTACTS AND LOCATIONS:
Overall Officials: Seda Ayaz Taş, Phd, Principal Investigator — Abant Izzet Baysal University
Locations (3):
- Turkey (Türkiye) (3):
  - Bolu Abant İzzet Baysal University, Bolu, Bolu
  - Düzce Gökkuşağı Özel Eğitim ve Rehabilitasyon Merkezi, Düzce, Düzce
  - Kdz. Ereğli Gökkuşağı Özel Eğitim ve Rehabilitasyon Merkezi, Ereğli, Zonguldak Province

IPD SHARING:
Plan to Share IPD: No